CLINICAL TRIAL: NCT04509102
Title: *Full Title of the Submission: Psychostimulant Augmentation of Repetitive TMS (rTMS) for the Treatment of Major Depressive Disorder: A Randomized, Placebo-controlled Clinical Trial
Brief Title: Psychostimulant Augmentation of Repetitive TMS for the Treatment of Major Depressive Disorder
Acronym: Stimulant-rTMS
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Scott A. Wilke, MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-000050
Record Dates: First submitted 2020-06-29; First posted 2020-08-11 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Disorder
Keywords: MDD, Randomized, rTMS; Randomized; rTMS
MeSH Terms: conditions — Depressive Disorder, Major | interventions — SLI381

STUDY DESIGN:
Intervention Model Description: i. Prior to initiation of any study activities, participants will be randomly assigned to one of two treatment conditions: Adderall XR (n=15) versus placebo (n=15). Randomization will be completed by a biostatistician from the UCLA Clinical and translational science institute (CTSI) statistics core, who will generate the randomization list with stratification and provide this list to the UCLA pharmacy.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Only the biostatistician conducting the randomization will know each participant's treatment condition (Adderall XR versus placebo) for the duration of the trial. Participants, psychiatrists, and technicians delivering rTMS and collecting assessments will be blinded to treatment condition (Adderall XR versus placebo). Active medication will be over-encapsulated by the UCLA Research Pharmacy to appear identical to placebo capsules. At the conclusion of all treatments, participants will be asked whether they believe they received Adderall XR release versus placebo. The blind will then be broken and participants may elect to continue medication management at the discretion of their personal psychiatrist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator): Subjects randomized to Adderall will take an tablet/capsule by mouth daily.
  Interventions: Drug: Adderall-XR
- Placebo (Placebo Comparator): Subjects randomized to placebo will take an identical-appearing tablet/capsule and, in order to maintain blinding, will also take one tablet by mouth daily. The placebo substance will be sugar.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Adderall-XR — Subjects randomized to Adderall XR will initiate treatment with 15 mg daily (one 15 mg tablet each morning) for 21 days.
  Arms: Active
Drug: Placebo — Subjects randomized to placebo will take an identical-appearing tablet/capsule and, in order to maintain blinding, will also take one tablet by mouth daily. The placebo substance will be sugar for 21 days.
  Arms: Placebo

SUMMARY:
This study analyzes the affects or Adderall extended-release (XR) in Subjects receiving brain stimulation therapy for the treatment of Major Depressive Disorder. Subjects will be assigned by chance to active or placebo group. Active group will be asked to take one 15 mg pill once daily of Adderall XR (amphetamine) and the Placebo group will be asked take an identical appearing tablet/capsule, one tablet by mouth daily. The placebo tablet has no active ingredients and has no affect on the body or mind. With the exception of the study drug, all other study activities between both groups will be identical. Subjects will use the assigned study drug two weeks before therapy and throughout the first 10 therapy treatments. A total of seven(7) visits will be required for screening, drug assignment, and completion of mood assessments. This study will enroll a total of 30 Subjects.

DETAILED DESCRIPTION:
This study aims to recruit 30 subjects between the ages of 18-65 who meet the Diagnostic and Statistical Manual of Mental Disorders (DSM-V) criteria for a current episode of major depressive disorder. Participants will be recruited from the population of patients seeking rTMS from the University of California Los Angeles(UCLA) Transcranial Magnetic Stimulation Clinic. All patients considered for participation in the study will carry a diagnosis of major depression as established by the referring psychiatrist and this will be confirmed based on an interview using the Mini International Neuropsychiatric Interview (MINI). Moreover, they will meet criteria for treatment resistance as defined by lack of response to two prior antidepressant trials at adequate dosage and duration. After providing voluntary, capable, informed consent, participants will be enrolled in the study. Participants will then complete baseline assessments including the Antidepressant Treatment History Form (ATHF) and the 30-item Inventory of Depressive Symptomatology Self Report (IDS-SR30) as well as the clinician-rated 17-item Hamilton Depression Rating Scale (HAM-D17).

Once a diagnosis of treatment resistant major depression has been established, the primary outcome measure will be the IDS-SR30 score, which is our standard procedure for monitoring treatment outcome in the TMS clinic. Participants will be randomly assigned to one of two treatment conditions: Adderall XR (n=15) versus placebo (n=15). Participants and all research team members will be blinded to the assigned treatment condition. Timing of all steps in the study protocol will use 'study time', meaning that although patients remain on the drug during weekends, only weekdays (Mon-Fri) count when assessing progress through the protocol. For example, a patient that started day 1 of the study on a Thursday, would reach day 5 on Wednesday the following week. Adderall XR or placebo will be initiated at least 10 days prior to the start of rTMS treatment in order to assess side effects and establish stable mood on the study drug. In order to study how Adderall XR affects response to rTMS, independent of any direct antidepressant effects, patients must exhibit stable mood prior to initiating rTMS. IDS-SR30 and HAM-D17 will be repeated on study days 5 and 10 on drug to determine if patients have a stable baseline mood (see study schedule chart, below). Patients will be considered to exhibit stable mood and qualify for initiating treatment if the IDS-SR30 score changes by less than 10% between assessments at study day 5 and 10.

The investigators predict that some patients may exhibit improvement in IDS score at day 5, however, if they exhibit significant additional improvement between day 5 and 10, starting rTMS will be delayed until depression scores are stabilized. Specifically, if the mood score changes by more than 10%, the Subject will wait an additional 5 days or multiples of 5 days up to 15 days as needed, until the weekly change in mood score meets this criterion. The investigators predict that few of these treatment-resistant, depressed patients will exhibit more than a couple weeks of continuous improvement, but if they do they may be better suited by continuing stimulant treatment with their primary provider rather than undergoing TMS. Study subjects who no longer complain of depression and no longer meet criteria for Major Depressive Disorder (MDD) after initiating treatment (Adderall XR vs. placebo) will be removed from the study because rTMS is no longer indicated. For such patients, the blind will be broken and they would have the option to continue the study medication at the discretion of their primary prescribing physician.

Participants will be assessed for medication side effects alongside IDS-SR30 assessments and rTMS will begin once they exhibit stably depressed mood. Participants in both treatment groups will begin a standard, FDA approved rTMS treatment protocol, delivered with a Magstim or Magventure device. Participants will be assessed for side effects at each rTMS treatment session. Participants will complete the IDS-SR30, HAM-D17 and a Visual Analog Scale (VAS) for overall tolerability after 5 and 10 rTMS treatment sessions. After completion of the 10th treatment session and the final set of assessments, all study related activities will be complete and the blind will be broken.

Based on our recent observational study, the investigators predict that the effect Adderall XR on rTMS outcome will be most apparent early in the treatment course. Moreover, in our standard treatment algorithm, rTMS treatment parameters are generally kept uniform during the first 10 treatments and begin to diverge thereafter depending on treatment response. Thus, examining outcomes after treatment 10 will yield the best controlled dataset for detecting a significant effect of the study drug. Patients may complete additional rTMS treatments at the discretion of the treating physician, and may elect to continue taking the study drug at the discretion of their prescribing psychiatrist. Therefore, patients that exhibit significant improvement in depression while taking Adderall XR would have the option to continue beyond the initial 10 treatments. Otherwise, patients will discontinue the study medication at this point and given the low dose and short duration of treatment, it is not anticipated that patients will require any need to wean off the study medication.

ELIGIBILITY:
Inclusion Criteria:

* All subjects will be between the ages of 18-65 and will meet DSM-V criteria for a current episode of major depressive disorder.
* Meet criteria for treatment resistance as defined by lack of response to two prior antidepressant trials at adequate dosage and duration. Participants may use any psychotropic medications other than psychostimulants or benzodiazepines, and may continue these medications during the study.
* The outside treating psychiatrist must agree that enrollment in the study is safe and acceptable for the subject.

Exclusion Criteria:

* Inability to give informed consent
* Lifetime diagnosis of bipolar affective disorder
* Lifetime diagnosis of major depressive disorder with psychotic features, schizophrenia, schizoaffective disorder, or any other psychotic disorder
* History of psychotic symptoms
* Lifetime diagnosis of substance use disorder
* History of stimulant misuse or abuse
* Active substance abuse
* Anxiety, tension, or agitation that is of sufficient severity to make it difficult for the subjects to tolerate psychostimulants and/or 10 Hz rTMS treatment
* Current use of psychostimulant medication
* Current use of benzodiazepines
* Current use of an Monoamine oxidase inhibitors (MAOI) or use of an MAOI within the past two weeks
* History of hypersensitivity to Adderall XR
* History of intolerance of any psychostimulant medication
* Pregnancy, breastfeeding, or plans to become pregnant during the study period
* Glaucoma
* Presence of motor tics or family history of tic disorder
* Symptomatic cardiovascular disease including hypertension, coronary artery disease, arteriosclerosis, cardiomyopathy, or arrhythmia
* Hyperthyroidism
* Structural cardiac abnormalities
* Family history of sudden cardiac death in a first degree relative
* History of epilepsy or seizure
* History of stroke
* History of brain tumor
* Presence of any metal in the head
* Presence of pacemaker or medical devices implanted close to the site of magnetic stimulation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Mean Percent Change in Self-rated Inventory of Depressive Symptoms | up to 4 weeks- 6 assessments from baseline to study completion
  Mean percent change in Self-rated Inventory of Depressive Symptoms assessment scores for subjects, compared between placebo and Adderall XR groups. The 30 item Inventory of Depressive Symptomatology (IDS) (Rush et al. 1986, 1996) assess the severity of depressive symptoms. It is a 30 -item questionnaire with scores ranging from 0-3 per time. Minimum and maximum values are 0 and 84, respectively. Higher score indicates a worsening in depressive symptoms and a lower score indicated an improvement in depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Wilke, MD, Principal Investigator — UCLA Semel
Locations (1):
- UCLA Semel, Los Angeles, California, United States